CLINICAL TRIAL: NCT05495828
Title: Observational Study of Orelabrutinib Therapy in Patients With Relapsed or Refractory B-cell Lymphoma Intolerant to Other Bruton Tyrosine Kinase Inhibitors
Brief Title: Orelabrutinib Therapy in Patients With r/r B-cell Lymphoma Intolerant to Other Bruton Tyrosine Kinase Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Other Study IDs: intolerant to BTK inhibitors
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — orelabrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orelabrutinib: Patients with relapsed or refractory B-cell lymphoma (including r/rCLL/SLL, r/rMCL) intolerant to ibrutinib/zanubrutinib or other BTK inhibitors who have decided to receive Orelabrutinib therapy
  Interventions: Drug: Orelabrutinib

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib, 150mg, po, qd
  Other Names: ICP-022

SUMMARY:
To evaluate the safety and effecacy of Orelabrutinib therapy in patients with relapsed or refractory B-cell lymphoma (including R /rCLL/SLL and R /rMCL) who are intolerant to ibrutinib/zanubrutinib or other BTK inhibitors

DETAILED DESCRIPTION:
The efficacy of first-generation BTKi ibrutinib in the treatment of B-cell lymphoma is reasonable, but the kinase selectivity is poor and the off-target effect is increased. It is associated with non-BTK-related adverse reactions such as bleeding, atrial fibrillation, diarrhea and rash.This is the reason why some patients stop taking BTKi and cannot benefit from long-term treatment. Orelabrutinib kinase is highly selective. The safety of the treatment of 266 Chinese patients with B-cell malignancies (including r/r CLL/SLL, r/r MCL, r/r WM, r/r MZL, r/r CNSL) showed that no ≥ grade 3 atrial fibrillation occurred.The incidence of grade 3 diarrhea and severe bleeding adverse events was lower than that of ibrutinib and zanubrutinib.Therefore, the aim of this study was to evaluate the safety and efficacy of self-selected switching to obrutinib in patients with relapsed or refractory B-cell lymphoma intolerant to ibrutinib/zanubrutinib therapy

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18 years, both sexes; 2) Confirmed by the following diagnostic criteria CLL/SLL: relapsed or refractory chronic lymphocytic leukemia/small lymphocytic lymphoma confirmed by flow cytometry or histopathology according to iwCLL2018 criteria MCL: Recurrent or refractory mantle cell lymphoma histopathologically confirmed: including cytogenetic testing T (11;14) Mantle cell lymphoma with positive/high immunohistochemical expression of Cyclin D1 3) Previous treatment with ibrutinib/zanubrutinib/or other BTK inhibitors and any of the following conditions were defined by the investigator as poor tolerance to ibrutinib/zanubrutinib or other BTK inhibitors: A) Grade ≥2 nonhematologic toxicity lasting >7 days with or without treatment; B) any non-hematological toxicity of ≥ grade 3 ; C) Grade 3 neutropenia with infection or fever; D) Grade 4 hematologic toxicity that persisted until the investigator chose to discontinue ibrutinib/ zanubrutinib or other BTK inhibitors due to toxicity rather than disease progression 4) The investigator-initiated treatment decision to use Orelabrutinib (before study enrollment); 5) Life expectancy ≥3 months; 6) The patient or his or her legal representative voluntarily signed written informed consent

Exclusion Criteria:

* 1) Richter conversion (CLL/SLL) or disease progression during treatment with ibrutinib/ zanubrutinib or other BTK inhibitors; 2) Past treatment with Orelabrutinib; 3) Absolute neutrophil ANC<0.75×109/L, platelet PLT<50×109/L; 4) Blood biochemistry: total bilirubin (TBIL) >2 times the upper limit of normal ULN (unless Gilbert syndrome is diagnosed), AST or ALT>2.5× ULN; Serum creatinine (Cr) >1.5×ULN 5) Coagulation function: INR and APTT ≤1.5 × ULN; 6) Grade 3 or 4 adverse events related to ongoing unresponded treatment with ibrutinib/ zanubrutinib or other BTK inhibitors 7) Participate in research projects that use interventions outside the scope of routine clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed or refractory B-cell lymphoma (including r/rCLL/SLL, r/rMCL) intolerant to ibrutinib/zanubrutinib or other BTK inhibitors who have decided to receive Orelabrutinib therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
the adverse events of Special interest | up to two years
  the adverse events of Special interest: Diarrhea, atrial fibrillation/flutter, rash

SECONDARY OUTCOMES:
ORR | up to two years
  The proportion of CR + PR in different B cell lymphoma subtype
DCR | up to two years
  The proportion of CR + PR+SD in different B cell lymphoma subtype
DOR | up to two years
  The time from the first remission to the first progression of the disease
PFS | up to two years
  The time from the start of medication to the first progression of disease or death
OS | up to two years
  The time from initiation of the drug to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Shenmiao Yang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Deparment of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No